CLINICAL TRIAL: NCT06711822
Title: Prospective, Multicenter, Single-group Clinical Trial Evaluating the Safety and Effectiveness of ShockPulse-10 in the Treatment of Coronary Artery Calcification
Brief Title: The Safety and Performence of ShockPulse-10 in Patients with Coronary Artery Calcification
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keya Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-27
Record Dates: First submitted 2024-11-20; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Coronary Arterial Disease (CAD); Calcification; Heart
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device (Experimental): Shockplus-10
  Interventions: Device: Shockplus-10

INTERVENTIONS:
Device: Shockplus-10 — Patients with coronary artery calcification who are planned to undergo PCI and are deemed in need of ShockPulse-10 treatment by their physicians

SUMMARY:
This study is an exploratory, multicenter, single-group clinical trial aimed to evaluate the clinical outcomes of using ShockPulse-10 in the treatment of coronary artery calcification .

DETAILED DESCRIPTION:
The study will be conducted at 8 sites in China and up to 205 participants will be followed for 180 days post procedure.

Patients ≥18 years of age scheduled for stent procedure with evidence of significant calcified stenosis of left main, or left anterior descending, right coronary artery or left circumflex will be eligible to enroll in the study. The primary endpoint of the study will evaluate procedure success,procedure success defined as successful stent implantation, residual stenosis degree ≤30% , and no major adverse cardiac events (MACE) occurring during hospitalization.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient is ≥ 18 years of age;
2. Patients with significant coronary artery disease (including stable or unstable angina and asymptomatic myocardial ischemia) who are suitable for PCI treatment;
3. A single newly developed stenosis of the target vessel, which is the left anterior descending artery, right coronary artery, or circumflex artery (or its branches), with stenosis degree ≥70% or ≥50% (Visually inspect ) and accompanied by evidence of ischemia;
4. The target lesion is a primary, in situ coronary artery lesion;
5. The reference vessel diameter for the target lesion is 2.0-4.0mm, and the length of the target lesion is ≤40mm (Visually inspect);
6. Visual assessment indicates that the lesion site can accommodate the passage of a pre-dilator or trial instrument through the lesion;
7. The target lesion site has moderate to severe calcification (meeting one of the following conditions)：

   ① Angiography: Moderate calcification :clearer and more easily visible high-density shadows during cardiac pulsation; Severe calcification :clear high-density shadows both during and at rest;

   ② IVUS calcium score ≥2 points for superficial intimal, deep medial, and mixed calcification;
8. TIMI grade 3 in target vessel before registration (pre-dilation is allowed);

Key exclusion Criteria:

1. Left ventricular ejection fraction < 40%；
2. NYHA class III or IV heart failure；
3. Patients with single coronary artery supply;
4. Patients with evidence of dissection at the site of the lesion on imaging;
5. The imaging suggests that the vascular pathway is tortuous, making it difficult for the pre-dilatation device to reach the target location or to be retrieved;
6. Patients with active systemic infections;
7. Patients with uncontrollable severe hypertension (systolic pressure > 180 mmHg or diastolic pressure > 110 mmHg);
8. Patients with coagulopathy, hypercoagulable state or significant bleeding tendency (hemoglobin <10g/dL or platelet count <80×10^9/L);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedure success | immediately post-procedure or prior to discharge, whichever comes first
  Procedure success defined as successful stent implantation, residual stenosis degree ≤30% , and no major adverse cardiac events (MACE) occurring during hospitalization
Freedom from major adverse cardiac events (MACE) within 30 days of the index procedure | 30（±7days）days post index procedure
  Freedom from major adverse cardiac events (MACE) within 30(±7days) days of the index procedure；MACE is defined as:Cardiac death; or Myocardial Infarction (MI): or Target Vessel Revascularization

CONTACTS AND LOCATIONS:
Overall Officials: XIANTAO SONG, Dortor, Principal Investigator — Beijing Anzhen Hosipital
Locations (1):
- Beijing Anzhen Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No